CLINICAL TRIAL: NCT06941493
Title: Effect of Normal Birth Simulation and Podcast Training Given to Pregnant Women on Birth Fear, Belief and Self-Efficacy: Randomized Controlled Study
Brief Title: Effect of Normal Birth Simulation and Podcast Training Given to Pregnant Women on Birth Fear, Belief and Self-Efficacy
Status: Not yet recruiting | Type: Observational
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Sema Göçmez, Lecturer, Eskisehir Osmangazi University
Other Study IDs: GO 2025/1004
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Fear of Childbirth; Childbirth Education
Keywords: Pregnancy; prenatal education; simulation; podcasd

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- simulation training group: Normal birth simulation training will be given to this group for an average of 1 hour for 4 weeks in the simulation laboratory of Bucak School of Health.
- podcast eğitim grubu: The podcast group will be sent a 20-minute podcast video in parallel with the simulation group for 4 weeks In the first session, the podcast file prepared by the researcher will be uploaded to the smartphones of the pregnant women and it will be checked that the file works smoothly. Pregnant women will be called in the relevant weeks to confirm whether they are watching the podcast and whether there are any problems.
- control group: No intervention will be made to the control group by the research team, this group will only complete the standard prenatal education process in the pregnant class.

SUMMARY:
According to the World Health Organization (WHO), health education is "educational practices carried out in order to provide individuals, families and society with a healthy lifestyle, to adopt and implement the measures to be taken to improve their health, to get them used to using the health services offered, to persuade them to improve their health and their environment, to make them reach a common decision and to direct them to action" . As in all stages of life, it is known that the trainings given during pregnancy contribute to the protection of maternal and infant health. The aim of childbirth preparation trainings given for a healthy pregnancy and birth process is to develop positive health behaviors in line with the needs of the person, to increase confidence in oneself and one's body, to reduce the stress caused by the fear and uncertainty associated with childbirth encoded since the past, to ensure the desire to give birth normally and to ensure secure mother-baby bonding. Although prenatal education has positive contributions to the pregnancy and birth process, it has been determined that the verbal expression of the teaching style of routine prenatal education leads to a passive acceptance without establishing a cause and effect relationship by weakening the learning effect and moving away from mutual interaction. In the study conducted by Downe et al. (2019), it was determined that routine prenatal education was insufficient to meet the information needs of women. It is thought that prenatal education prepared through simulation and podcast by utilizing the advantages of digital technology on health education can be useful in increasing women's beliefs and self- efficacy towards normal delivery, reducing their fear of childbirth, increasing their knowledge levels and eliminating misinformation. From this point of view, our study is aimed to bring innovation to the literature. The aim of this study is to examine the effect of simulation and podcast education used in prenatal education on pregnant women's fear of childbirth, birth beliefs and birth self-efficacy.

he main questions it aims to answer are

Research question 1: Do the trainings given to pregnant women affect fear of childbirth? Research question 2: Do the trainings given to pregnant women affect birth self-efficacy? Research question 3: Does education for pregnant women affect birth beliefs? To see if the drug ABC treats severe asthma, the researchers will compare it to a placebo (a substance that looks like a drug, but does not contain one).

To assess the effectiveness of prenatal education, the researchers will Group 1 will be trained with simulated labor for 4 weeks in addition to routine pregnancy education Group 2 will be shown podcast videos simulating childbirth for 4 weeks in addition to routine pregnancy education Group 3 will be provided with routine prenatal education

ELIGIBILITY:
Inclusion criteria Able to speak, understand and write Turkish,

* Those between the ages of 18-35
* Spontaneous pregnancy,
* Primiparous pregnant women
* 30-34. week of pregnancy
* Any health problems (hypertension, heart, diabetes, tuberculosis, HIV, cancer, etc.) non-
* Singleton pregnancy
* Participating in routine pregnancy education class
* Having a phone with internet connection for training meetings Exclusion criteria from the study
* Pregnant women diagnosed with medium and high risk pregnancy (such as oligohydramnios, preeclampsia, heart disease, diabetes, placenta previa)
* Presence of any diagnosed psychiatric disease (such as anxiety, depression)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Woman
Study Population: Healthy pregnant women aged 18-35 years, planning to give birth normally and participating in prenatal education programs
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2025-05-16 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Wijma Birth Expectancy/Expectation Questionnaire (W-DEQ) A Version | 30-34 weeks of gestation
  The "Wijma Birth Expectancy/Expectation Scale A Version (W-DEQ A)" developed by K. Wijma et al. in Sweden in 1998 was adapted into Turkish by Körükçü et al. in 2012. The W-DEQ consists of 33 items and is a six-point Likert-type scale. Item responses are numbered from 0 to 5, with 0 indicating "completely" and 5 indicating "not at all". The minimum score is 0 and the maximum score is 165. The cut-off value is 85 points and a score of 85 and above is expressed as clinical fear. A high total score means that the degree of fear experienced is also high.
  W-DEQ score ≤ 37 mildly,
  * W-DEQ score = 38-65 moderate,
  * W-DEQ score = 66-84 in severe degree,
  * W-DEQ score ≥ 85 indicates a clinical degree of fear. Questions 2, 3, 6, 7, 7, 8, 11, 12, 15, 19, 20, 24, 25, 27 and 31 in the scale are negatively loaded and are calculated by inverting them in the opposite direction in order to ensure compliance in the measurement. The cronbach alpha value of the scale was found to be 0.89

IPD SHARING:
Plan to Share IPD: Yes